CLINICAL TRIAL: NCT01614912
Title: Long-term Extension Study of SM-13496 (Lurasidone HCl) in Patients With Schizophrenia <Phase 3>
Brief Title: Long-term Extension Study of SM-13496 (Lurasidone HCl) in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1001057; JapicCTI-121860 (Registry Identifier: JAPIC Clinical Traials Information)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SM-13496 (Experimental)
  Interventions: Drug: SM-13496

INTERVENTIONS:
Drug: SM-13496 — 40 or 80 mg once daily orally

SUMMARY:
The study evaluates the long term safety and efficacy of SM-13496 in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are considered by the investigator eligible for the present study with no significant safety concerns
* Patients who are fully informed of and understand the objectives, procedures, and possible benefits and risks of the study and who provide written voluntarily consent to participate in the study

Exclusion Criteria:

* Patients who are planning pregnancy for the expected duration of the study
* Patients who are otherwise considered ineligible for the study by the investigator

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- 69 Sites, Tokyo, Etc, Japan
- 10 Sites, Kuala Lumpur, Etc, Malaysia
- 22 Sites, Seoul, Etc, South Korea
- 14Sites, Taipei, Etc, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group: SM-13496 40 mg or 80 mg was orally administered for 26 weeks to the participants who completed the prior study (D1001056), in which, SM-13496 (40 mg or 80 mg) or placebo was administered for 6 weeks.
Period: Overall Study
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Started | 284
Completed | 159
Not Completed | 125

BASELINE CHARACTERISTICS:
Population: ITT (intent-to-treat) population
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 152
Region of Enrollment [Number; unit: participants]
  Japan | 126
  Taiwan | 39
  Korea, Republic of | 76
  Malaysia | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at LOCF Endpoint
Description: The PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items and three subscales: the Positive subscale contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility; the Negative subscale contains seven questions to assess blunted effect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of motivation, and similar symptoms; and the General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity.
Time Frame: DB baseline and up to 32 weeks (LOCF endpoint)
Population: ITT (intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 281
units on a scale | -28.4 (22.2)

2. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity of Illness (CGI-S) Score at LOCF Endpoint
Description: CGI-S is a clinician-rated assessment of the participant's current disease state on a 7-point scale, where a higher score is associated with greater severity of the disease.
  Baseline in the prior study (D1001056, double-blind [DB] baseline) was defined as baseline of the prior study. Baseline in the present study (D1001057, extension [EXT] baseline) was defined as Week 6 in the prior study.
  The last post-baseline visit data collected during the study treatment of the present study were carried forward and defined as the last observation carried forward (LOCF) endpoint.
Time Frame: DB baseline and up to 32 weeks (LOCF endpoint)
Population: ITT (intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 281
units on a scale | -1.46 (1.36)

3. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score at LOCF Endpoint
Description: The PANSS is comprised of 30 items and three subscales. The Positive subscale contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS Positive subscale score is the sum of all 7 items and ranges from 7 through 49. A higher score is associated with greater illness severity.
Time Frame: DB baseline and up to 32 weeks (LOCF endpoint)
Population: ITT (intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 281
units on a scale | -8.4 (6.8)

4. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score at LOCF Endpoint
Description: The PANSS is comprised of 30 items and three subscales. The Negative subscale contains seven questions to assess blunted effect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of motivation, and similar symptoms. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS Negative subscale score is the sum of all 7 items and ranges from 7 through 49. A higher score is associated with greater illness severity.
Time Frame: DB baseline and up to 32 weeks (LOCF endpoint)
Population: ITT (intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 281
units on a scale | -6.9 (5.9)

5. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscale Score at LOCF Endpoint
Description: The PANSS is comprised of 30 items and three subscales. The General Psychopathology subscale addresses other 16 symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS General Psychopathology subscale score is the sum of all 16 items and ranges from 16 through 112. A higher score is associated with greater illness severity.
Time Frame: DB baseline and up to 32 weeks (LOCF endpoint)
Population: ITT (intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 281
units on a scale | -13.1 (11.7)

6. Secondary Outcome: Proportion of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Proportion of participants with treatment-emergent adverse events. An adverse event was defined as any untoward medical occurrence in a patient treated with a medicinal (investigational) product and which did not necessarily have a causal relationship with this treatment. Treatment-emergent adverse events are defined as adverse events with a start date on or after the date of initial administration of study drug in the present study through the end of follow-up or adverse events occurring before the date of initial administration of study drug in the present study and worsening during the study treatment in the present study.
Time Frame: EXT baseline and up to 26 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 282
Participants | 215

7. Secondary Outcome: Proportion of Participants With TEAEs Leading to Discontinuation
Time Frame: EXT baseline and up to 26 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 282
Participants | 39

8. Secondary Outcome: Proportion of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: Proportion of participants with treatment-emergent adverse events. A serious adverse event was defined as an AE that met one or more of the following criteria: Resulted in death; Was life-threatening (i.e., a patient was at immediate risk of death at the time of the event, not an event where occurrence in a more severe form might have caused death); Required hospitalization or prolongation of existing hospitalization; Resulted in persistent or significant disability or incapacity; Was a congenital anomaly or birth defect; Was an important medical event that might jeopardize the patient or might require medical intervention to prevent one of the outcomes listed above.
Time Frame: EXT baseline and up to 26 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
Number analyzed (Participants) | 282
Participants | 31

ADVERSE EVENTS:
Time Frame: EXT baseline and up to 24 weeks
Description: Baseline in the present study (D1001057, extension [EXT] baseline) was defined as Week 6 in the prior study (D1001056). Both TEAEs and treatment-emergent serious adverse events are presented for the safety population defined as subjects who receive at least one of the study drug.
  Patients experiencing multiple adverse events are counted once in each category.
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group
All-Cause Mortality (participants affected / at risk) | 1/282
Serious Adverse Events (participants affected / at risk) | 31/282
Other Adverse Events (participants affected / at risk) | 184/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group (N=282)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Diabetes insipidus (Endocrine disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Blood hyposmosis (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Convulsion (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 17
Renal failure acute (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SM-13496 (Lurasidone HCl) 40-mg or 80-mg Group (N=282)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Long QT syndrome (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 2
Hyperprolactinaemia (Endocrine disorders) | 1
Vision blurred (Eye disorders) | 3
Conjunctivitis (Eye disorders) | 2
Chalazion (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Eye discharge (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Posterior capsule opacification (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 5
Salivary hypersecretion (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Periodontitis (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 3
Oedema peripheral (General disorders) | 3
Chest discomfort (General disorders) | 2
Gait disturbance (General disorders) | 2
Pyrexia (General disorders) | 2
Drug ineffective (General disorders) | 1
Fatigue (General disorders) | 1
Irritability (General disorders) | 1
Malaise (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Nasopharyngitis (Infections and infestations) | 30
Upper respiratory tract infection (Infections and infestations) | 14
Influenza (Infections and infestations) | 5
Hordeolum (Infections and infestations) | 3
Tinea pedis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Acarodermatitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Carbuncle (Infections and infestations) | 1
Dermatophytosis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Genital infection fungal (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Pyoderma (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sweating fever (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 4
Road traffic accident (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Blood prolactin increased (Investigations) | 9
Weight increased (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 2
Blood uric acid increased (Investigations) | 2
Protein urine present (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Abnormal weight gain (Metabolism and nutrition disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Akathisia (Nervous system disorders) | 31
Headache (Nervous system disorders) | 15
Tremor (Nervous system disorders) | 10
Dyskinesia (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 6
Dystonia (Nervous system disorders) | 5
Bradykinesia (Nervous system disorders) | 3
Cervicobrachial syndrome (Nervous system disorders) | 1
Drooling (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dyslalia (Nervous system disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Hyperaesthesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Oromandibular dystonia (Nervous system disorders) | 1
Parkinsonian gait (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Poor quality sleep (Nervous system disorders) | 1
Tardive dyskinesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 32
Schizophrenia (Psychiatric disorders) | 10
Anxiety (Psychiatric disorders) | 23
Psychotic disorder (Psychiatric disorders) | 4
Agitation (Psychiatric disorders) | 5
Aggression (Psychiatric disorders) | 2
Depressed mood (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 2
Abulia (Psychiatric disorders) | 1
Impulsive behaviour (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Persecutory delusion (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2
Balanitis (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 8
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 6
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 2
Dental care (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Somnolence (Nervous system disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes